CLINICAL TRIAL: NCT04533074
Title: Microbiological Evaluation of Single Versus Multiple Visits Regeneration Using MALDI-TOF Mass Spectrometry (A Randomized Controlled Clinical Trial)
Brief Title: Microbiological Evaluation of Single Versus Multiple Visits Regeneration Using MALDI-TOF Mass Spectrometry
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to the COVID-19 pandemic
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MALDI-TOF MS regeneration
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Pulp Necroses; Tooth, Nonvital
MeSH Terms: conditions — Dental Pulp Necrosis; Tooth, Nonvital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-visit regeneration protocol (Experimental)
  Interventions: Biological: Single-visit regeneration protocol
- Multiple-visits regeneration protocol (Active Comparator)
  Interventions: Biological: Multiple-visits regeneration protocol

INTERVENTIONS:
Biological: Single-visit regeneration protocol — In a single visit, access opening, minimal instrumentation and irrigation will be done. After irrigation and drying, the apical tissue will be irritated to evoke bleeding in the canal, using a precurved K-file 2mm past the apical foramen, with the goal of having the entire canal filled with blood to the level of the cemento-enamel junction. The bleeding will be stopped at a level that allows for 3-4 mm of restorative material. Three millimeters of Biodentine will then be placed directly over the blood clot of each tooth. A 3-4 mm layer of glass ionomer is flowed gently over the capping material. Each access cavity will be restored using composite resin.
  Arms: Single-visit regeneration protocol
Biological: Multiple-visits regeneration protocol — In the first visit, access opening, minimal instrumentation and irrigation will be done. The root canal will be then dried and filled with calcium hydroxide paste. The tooth will be sealed with an intermediate restorative material (IRM), and the patient will be dismissed for 1-4weeks. In the second appointment, response to initial treatment will be assessed and the steps will be repeated if symptoms are persistent. If there are no symptoms, evoking bleeding to the level of the cemento-enamel junction will be done followed by Biodentine application over the blood clot with final glass ionomer and composite restorations.
  Arms: Multiple-visits regeneration protocol

SUMMARY:
Aim of the study is to assess canal disinfection using matrix assisted laser desorption ionization-time of flight mass spectrometry (MALDI-TOF MS) in single visit and multiple visit regeneration protocols, and to assess clinical and radiographic outcomes of single visit and multiple visit regeneration protocols.

DETAILED DESCRIPTION:
Thirty patients with necrotic immature permanent teeth showing periapical lesions will be randomly divided in two groups: group (1) single visit regeneration and group (2) multiple visits regeneration protocol, in which calcium hydroxide will be applied for one week or more according to resolution of signs and symptoms. Dentin debris collected on a file will be taken as microbiologic sample to be cultured and examined by MALDI-TOF MS. This will be performed after the access cavity preparation and after irrigation in both groups, these samples will be labelled A and B, respectively. In group (2) there will be a third sample labeled C which will be taken after the removal of the intra canal calcium hydroxide.

ELIGIBILITY:
Inclusion Criteria:

* Immature permanent upper anterior teeth.
* Necrotic teeth confirmed by sensibility test.
* Teeth with periapical lesions confirmed by periapical radiograph using paralleling device.

Exclusion Criteria:

* Teeth with orthodontic wires or brackets.
* Patient with history of allergy to any medication.
* Patient with history of bleeding disorders.
* Patient with medical illness or taking medications.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Microbiological assessment | 24 hours
  The presence or absence of reduction in types of micro-organisms in root canals
Tooth vitality | up to 12 months
  Tooth vitality will be assessed by sensibility testing using thermal stimulation, binary (yes or no).
Tooth mobility | up to 12 months
  4. Mobility will be recorded according to Grace & Smales Mobility Index
  * Grade 0: No apparent mobility
  * Grade 1: Perceptible mobility <1mm in buccolingual direction
  * Grade 2: 1mm< but <2mm
  * Grade 3: 2mm< or depressibility in the socket
Healing of periapical lesions | up to 12 months
  Periapical index score (PAI) will be used for identification of apical periodontitis on both periapical radiography and Cone-beam computed tomographic (CBCT).
  It is a 6-point (0 -5) scoring system with 2 additional variables, expansion of cortical bone and destruction of cortical bone.The PAI will be determined by the largest extension of the lesion on periapical radiography and CBCT scans in 3 dimensions: axial, sagittal, and coronal.
  * Score 0 Intact periapical bone structures.
  * Score 1 Diameter of periapical radiolucency "0.5-1 mm.
  * Score 2 Diameter of periapical radiolucency "1-2 mm.
  * Score 3 Diameter of periapical radiolucency "2-4 mm.
  * Score 4 Diameter of periapical radiolucency "4-8 mm.
  * Score 5 Diameter of periapical radiolucency "8 mm.
  * Score (n)# E: Expansion of periapical cortical bone.
  * Score (n)# D: Destruction of periapical cortical bone.
Root lengthening | up to 12 months
  The root length will be measured as a straight line from the CEJ to the radiographic apex of the tooth. This will be measured on both periapical radiography and Cone-beam computed tomographic (CBCT) in millimeters.
Root thickening | up to 12 months
  The dentinal wall thickness for both the preoperative and recall images will be measured at the level of the apical one third of the preoperative root canal length measured from the CEJ. The root canal width and the pulp space will be measured at this level, and the remaining dentin thickness will be calculated by subtracting the pulp space from the root canal width.

CONTACTS AND LOCATIONS:
Overall Officials: Pervine H. Sharaf, M.Sc, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Raef A Sherif, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Ashraf M Zaazou, PhD, Study Chair — Faculty of Dentistry, Alexandria University, Egypt; Rania M ElBackly, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Garcia-Godoy F, Murray PE. Recommendations for using regenerative endodontic procedures in permanent immature traumatized teeth. Dent Traumatol. 2012 Feb;28(1):33-41. doi: 10.1111/j.1600-9657.2011.01044.x. Epub 2011 Jul 27. PMID 21794081
- [Background] El Ashiry EA, Farsi NM, Abuzeid ST, El Ashiry MM, Bahammam HA. Dental Pulp Revascularization of Necrotic Permanent Teeth with Immature Apices. J Clin Pediatr Dent. 2016;40(5):361-6. doi: 10.17796/1053-4628-40.5.361. PMID 27617376
- [Background] Diogenes A, Ruparel NB, Shiloah Y, Hargreaves KM. Regenerative endodontics: A way forward. J Am Dent Assoc. 2016 May;147(5):372-80. doi: 10.1016/j.adaj.2016.01.009. Epub 2016 Mar 24. PMID 27017182
- [Background] Flanagan TA. What can cause the pulps of immature, permanent teeth with open apices to become necrotic and what treatment options are available for these teeth. Aust Endod J. 2014 Dec;40(3):95-100. doi: 10.1111/aej.12087. PMID 25470507
- [Background] Aggarwal V, Miglani S, Singla M. Conventional apexification and revascularization induced maturogenesis of two non-vital, immature teeth in same patient: 24 months follow up of a case. J Conserv Dent. 2012 Jan;15(1):68-72. doi: 10.4103/0972-0707.92610. PMID 22368339
- [Background] Altaii M, Richards L, Rossi-Fedele G. Histological assessment of regenerative endodontic treatment in animal studies with different scaffolds: A systematic review. Dent Traumatol. 2017 Aug;33(4):235-244. doi: 10.1111/edt.12338. Epub 2017 Apr 20. PMID 28342218
- [Background] Saoud TMA, Ricucci D, Lin LM, Gaengler P. Regeneration and Repair in Endodontics-A Special Issue of the Regenerative Endodontics-A New Era in Clinical Endodontics. Dent J (Basel). 2016 Feb 27;4(1):3. doi: 10.3390/dj4010003. PMID 29563445
- [Background] McTigue DJ, Subramanian K, Kumar A. Case series: management of immature permanent teeth with pulpal necrosis: a case series. Pediatr Dent. 2013 Jan-Feb;35(1):55-60. PMID 23635900
- [Background] Khoshkhounejad M, Shokouhinejad N, Pirmoazen S. Regenerative Endodontic Treatment: Report of Two Cases with Different Clinical Management and Outcomes. J Dent (Tehran). 2015 Jun;12(6):460-8. PMID 26884781
- [Background] Chaniotis A. The use of a single-step regenerative approach for the treatment of a replanted mandibular central incisor with severe resorption. Int Endod J. 2016 Aug;49(8):802-12. doi: 10.1111/iej.12515. Epub 2015 Aug 21. PMID 26197881
- [Background] Nagata JY, Rocha-Lima TF, Gomes BP, Ferraz CC, Zaia AA, Souza-Filho FJ, De Jesus-Soares A. Pulp revascularization for immature replanted teeth: a case report. Aust Dent J. 2015 Sep;60(3):416-20. doi: 10.1111/adj.12342. Epub 2015 Jul 29. PMID 26219350
- [Background] Saoud TM, Huang GT, Gibbs JL, Sigurdsson A, Lin LM. Management of Teeth with Persistent Apical Periodontitis after Root Canal Treatment Using Regenerative Endodontic Therapy. J Endod. 2015 Oct;41(10):1743-8. doi: 10.1016/j.joen.2015.07.004. Epub 2015 Aug 14. PMID 26279479
- [Background] Jung IY, Lee SJ, Hargreaves KM. Biologically based treatment of immature permanent teeth with pulpal necrosis: a case series. J Endod. 2008 Jul;34(7):876-87. doi: 10.1016/j.joen.2008.03.023. Epub 2008 May 16. PMID 18571000
- [Background] Chueh LH, Ho YC, Kuo TC, Lai WH, Chen YH, Chiang CP. Regenerative endodontic treatment for necrotic immature permanent teeth. J Endod. 2009 Feb;35(2):160-4. doi: 10.1016/j.joen.2008.10.019. Epub 2008 Dec 12. PMID 19166764
- [Background] Tagelsir A, Yassen GH, Gomez GF, Gregory RL. Effect of Antimicrobials Used in Regenerative Endodontic Procedures on 3-week-old Enterococcus faecalis Biofilm. J Endod. 2016 Feb;42(2):258-62. doi: 10.1016/j.joen.2015.09.023. Epub 2015 Nov 11. PMID 26577870
- [Background] Topcuoglu G, Topcuoglu HS. Regenerative Endodontic Therapy in a Single Visit Using Platelet-rich Plasma and Biodentine in Necrotic and Asymptomatic Immature Molar Teeth: A Report of 3 Cases. J Endod. 2016 Sep;42(9):1344-6. doi: 10.1016/j.joen.2016.06.005. Epub 2016 Jul 15. PMID 27427186
- [Background] McCabe P. Revascularization of an immature tooth with apical periodontitis using a single visit protocol: a case report. Int Endod J. 2015 May;48(5):484-97. doi: 10.1111/iej.12344. Epub 2014 Aug 27. PMID 25066513
- [Background] Estrela C, Bueno MR, Azevedo BC, Azevedo JR, Pecora JD. A new periapical index based on cone beam computed tomography. J Endod. 2008 Nov;34(11):1325-1331. doi: 10.1016/j.joen.2008.08.013. Epub 2008 Sep 17. PMID 18928840